CLINICAL TRIAL: NCT05640544
Title: Gamma Entrainment Improve the Recovery of Awareness in Disorders of Consciousness
Brief Title: Gamma Entrainment Improve the Recovery of Awareness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20212209
Record Dates: First submitted 2022-10-31; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2021-12

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Sound

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sound and light stimulation in Gamma band (Experimental)
  Interventions: Other: Sound and light stimulation in Gamma band

INTERVENTIONS:
Other: Sound and light stimulation in Gamma band — We expect to screen out the efficacy of Gamma band in the prognosis and treatment of disorders of consciousness by various frequencies of stimulation.
  Optical stimulation:
  A computer program is used to control the flashing frequency of LED lights for stimulation. The serial port can convert the parallel data characters of the computer CPU into a continuous serial data stream. According to the frequency designed by experiment (10Hz, 20hz, 40hz, 80hz), we modulate the flicker frequency of LED lamp. LED lamp uses T8 lamp, diameter 25.4 mm, length 620 mm, and power 20W.
  Acoustic stimulation:
  We use Adobe Audition CC 2022 to modulate the tones. The tones modulated to 10Hz, 20Hz, 40Hz and 80Hz are play by noise-canceling headphones to the patients.

SUMMARY:
The purpose of this study is to elucidate the occurrence of Gamma entrainment and optimize the acousto-optic stimulation parameters to induce it in patients with disorders of consciousness (DOC), to explore the prognostic value of gamma entrainment in patients with DOC, and to clarify the effect of gamma entrainment on the recovery of awareness in DOC patients. This study is divided into three parts. The first and third parts are prospective cohort studies, the second part is a randomized cross control study. We recruit DOC patients, including vegetative state/unresponsive wakefulness syndrome (VS/UWS) or minimally conscious state (MCS). The patients receive sound and light stimulation in the Gamma band, and the changes of EEG are observed simultaneously to explore the occurrence of Gamma entrainment. Meanwhile, the changes of clinical behavior of patients before and after stimulation are evaluated.

ELIGIBILITY:
Inclusion Criteria:

Age 16-80 years; Clinical diagnosis of VS/UWS or MCS according to the CRS-R score within one week after admission; Time post-onset > 28 days.

Exclusion Criteria:

Previous history of acquired brain injury or psychiatric or neurodegenerative diseases; Clinical diagnosis of epilepsy; Visual or auditory pathway damage; Life threatening comorbidity, coexisting neoplasms, severe organ dysfunction, or unstable clinical condition (e.g., hemodynamic instability or severe respiratory failure); Incomplete clinical data.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes of EEG during stimulation procedure | Synchronous recording during stimulation procedure
  The changes of Gamma oscillation, the temporal and spatial distribution of Gamma band power and the changes of Gamma band brain network are analyzed before and after stimulation.

SECONDARY OUTCOMES:
CRS-R scale | at two weeks, 3 months, 6 months and 1 year after the onset.
  The CRS-R is used to assess patients with disorders of consciousness. The lowest score on each sub-scale represents reflexive activity; the highest represents behaviors mediated by cognitive input. The total score ranges between 0 (worst) and 23 (best).
Glasgow Outcome Scale - Extended (GOS-E) | at two weeks, 3 months, 6 months and 1 year after the onset.
  The GOS-E is one of the most widely used outcome instruments to assess global disability and recovery after brain injury. The Scale extends the original 5 GOS categories to 8. The total score ranges between 1 (worst) and 8 (best).
Modified Rankin Scale (mRS) | at two weeks, 3 months, 6 months and 1 year after the onset.
  The mRS assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. It is an ordered scale coded from 0 (no symptoms at all) to 6 (death).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Xijing Hospital, Air Force Medical University, Xi'an, China